CLINICAL TRIAL: NCT05296096
Title: PRotein Optimization With eXercise to Improve MUscle Mass and Functional outcomeS - a Pilot Feasibility, Randomized Controlled Trial
Brief Title: PRotein Optimization With eXercise to Improve MUscle Mass and Functional outcomeS
Acronym: PROXIMUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Nilesh M. Mehta, Faculty, Critical Care; Professor of Anesthesia, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: P00040737
Record Dates: First submitted 2022-03-08; First posted 2022-03-25 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Muscle Loss; Protein; Mobility; Pediatric ALL
Keywords: protein; exercise; mechanical ventilation; outcome; nutrition
MeSH Terms: conditions — Muscular Atrophy; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard protein and exercise (Active Comparator): All enrolled patients randomized to this arm will receive a baseline nutrition and nurse-driven mobility pathway and other evidence-based bundled strategies as standard of care.
  Interventions: Other: Protein dosage and rehabilitation team delivered exercise prescription
- High protein plus exercise (Experimental): High protein nutrition: To achieve the prescribed age-appropriate high protein target, dietitians will use EN preferentially, or if EN is contraindicated, PN may be used. High-protein EN formulas and/or protein supplements (powder or liquid) will be added to formula/breast milk feedings or administered separately in divided bolus doses. Dietitians routinely employ and customize these solutions in their scope of practice. When EN is insufficient to meet protein targets, PN may be prescribed to make up the deficit on or after the end of PICU day 3. Energy and protein delivery adequacy (% of prescribed goal) will be monitored daily by the study team.
  Patients in this arm will also be prescribed the age-appropriate highest-level of mobility by the rehabilitation team with a goal of 30 minutes duration, twice daily.
  Interventions: Other: Protein dosage and rehabilitation team delivered exercise prescription

INTERVENTIONS:
Other: Protein dosage and rehabilitation team delivered exercise prescription — The dietitian and rehabilitation team will be consulted on enrollment and will assess the patient for nutritional and functional status using the institutional criteria and physical exam. The study dietitian will prescribe the protein goal based on the randomization assignment and age group. For the high protein arm, protein goals will be 3g/kg/day for ages 1-1yrs, and 2.4g/kg/day for ages greater than 12 years.
  The rehabilitation team will determine the appropriate highest level of mobility (HLM) for the day in collaboration with the medical team on morning rounds. The rehabilitation team will prescribe passive or active participation in two 30-minute HLM sessions, individualized to their baseline function and clinical status and/or restrictions.

SUMMARY:
The investigators have designed a 2-center, pilot feasibility, randomized controlled trial (PROXIMUS) to determine the feasibility and safety of a larger multi center, randomized open-label trial comparing high protein combined with individualized exercise vs. standard management during the acute phase of critical illness in children. The investigators aim to determine the impact of the intervention on preservation of muscle mass; and functional status at 1 month and 6 months after randomization.

DETAILED DESCRIPTION:
Mortality in U.S. pediatric intensive care units (PICUs) is improving, resulting in an increased focus on the quality of life of survivors who often have persistent physical, cognitive, and psychological impairments. Mechanically ventilated children in particular experience immobilization and poor nutrient intake, which results in muscle loss during acute illness. Early mobility and optimal nutrition during acute critical illness have been associated with muscle mass preservation and decreased duration of mechanical ventilation. These interventions may have the potential to decrease preventable PICU-acquired morbidities. However, the optimal doses and long-term benefits of these interventions have not been shown in randomized studies of critically ill PICU patients.

Thus, the investigators will test the first pediatric-specific, inter-professional intervention that integrates high protein and individualized exercise. This intervention was developed by a team of experts in the fields of nutrition, early mobility, rehabilitative exercise, muscle ultrasound (US), and functional outcomes.

The investigators propose a 2-center, pilot feasibility, randomized controlled trial (PROXIMUS) with the following Specific Aims:

1. To determine the feasibility and safety of a randomized open-label trial comparing high protein combined with individualized exercise vs. standard management during the acute phase of critical illness in children;
2. To determine the impact of high protein and individualized exercise on preservation of muscle mass; and
3. To determine the impact of high protein and individualized exercise on functional status at 1 month and 6 months after randomization.

Outcomes: The investigators will assess feasibility with a composite measure that combines predetermined thresholds for screening, enrollment, allocation, and compliance/adherence with significant separation in doses of protein and exercise between the two arms. Safety will be defined as absence of difference in rates of new renal injury and exercise related adverse events.

Preservation of muscle mass will be assessed by percent daily change in US-measured quadriceps femoris muscle thickness (QFMT) during the PICU stay. The investigators will use a validated imaging protocol with high reliability and reproducibility. The investigators will also examine the difference in the normative standard scores (T-scores) between the two arms for the Pediatric Evaluation of Disability Inventory - Computer Adaptive Test (PEDI-CAT) assessment. Other secondary outcomes are Functional Status Scale, PedsQL, and muscle quality by US.

The investigators hypothesize that a larger trial will be feasible and safe. Patients randomized to the combined intervention will have lower decline in QFMT and better scores on PEDI-CAT assessment.

If proven feasible and safe, the PROXIMUS intervention has potential to profoundly change medical care in the PICU and substantially impact public health by improving long-term outcomes for the growing number of pediatric survivors of critical illness.

ELIGIBILITY:
Inclusion Criteria:

1. ICU patients aged 1 year (corrected) to <18 years
2. Require mechanical ventilation (endotracheal intubation or tracheostomy, or initiation of noninvasive ventilation) in the first 72 hours of PICU admission.
3. Able to consent to participate within 72 hours of initiation of mechanical ventilation initiation.

Exclusion Criteria:

* Patients unable to receive EN, PN, or who are on a specialized diet incompatible with the study intervention
* Fulminant liver failure
* Kidney failure (≥KDIGO Stage 3) without replacement therapy
* Functional Status Scale score at PICU admission <9
* End of life/redirection of care
* ECMO therapy
* Continuous neuromuscular blockade and/or bedrest is medically or surgically necessitated Participation in a conflicting interventional trial
* High risk of refeeding syndrome
* Inborn errors of metabolism
* High BSA burns.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of recruitment and adherence to study procedures | Through study completion, up to 10 days
  Feasibility (primary composite outcome) will be assessed by the following metrics: (1) >80% of eligible patients are approached for consent; (2) >35% of eligible patients are randomized (enrollment and consent); (3) >80% of consented patients receive study treatments (allocation and adherence).
Tolerability of protein intervention (serum creatinine change) | Through study completion, up to 10 days
  Incidence of treatment-related adverse events as assessed by 3-fold rise in serum creatinine or intolerance (new emesis or diarrhea) related to the study diet.
Safety of protein (new renal injury) and exercise interventions (any associated adverse events) | Through study completion, up to 10 days
  Incidence of treatment-related adverse events; specifically new renal injury or injury/discomfort associated with exercise.

SECONDARY OUTCOMES:
Change in Muscle mass thickness | Through study completion, up to 10 days
  As assessed by the change in quadriceps femoris (QF) muscle thickness between baseline measurement and measurement on study completion.
Functional assessment - motor, cognitive and responsibility | 6 months
  The investigators will administer the Pediatric Evaluation of Disability Inventory - Computer Adaptive Test (PEDI-CAT) test at 1 and 6 months after enrollment, and compare the scaled T-scores between the two trial arms at each time point. Higher score is better.
Multidimensional Pediatric Health related Quality of Life assessment (Physical, Emotional, Social, School Functioning domains) using a validated tool | 6 months
  The investigators will administer the Pediatric Health Related Quality of Life Questionnaire (PedsQoL) test at 1 and 6 months after enrollment, and compare the score between the two trial arms at each time point. Higher score on the developmentally appropriate questionnaire is better.
Assessment of Functional status - sensory, communication, motor, sensory and feeding | 6 months
  The investigators will administer the Functional Status Scale (FSS) assessment at 1 and 6 months after enrollment, and compare this scale between the two trial arms at each time point. The scale ranges from 6 to 30 points, lower is better,

OTHER OUTCOMES:
Protein catabolism (breakdown) | 10 days
  Proteomic profile measured in urine during the PICU stay

CONTACTS AND LOCATIONS:
Overall Officials: Nilesh Mehta, MD, Principal Investigator — Faculty, Boston Children's Hospital; Sapna R Kudchadkar, MD, PhD, Principal Investigator — Faculty, Johns Hopkins
Locations (2):
- United States (2):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mehta NM, Bechard LJ, Cahill N, Wang M, Day A, Duggan CP, Heyland DK. Nutritional practices and their relationship to clinical outcomes in critically ill children--an international multicenter cohort study*. Crit Care Med. 2012 Jul;40(7):2204-11. doi: 10.1097/CCM.0b013e31824e18a8. PMID 22564954
- [Background] Hauschild DB, Oliveira LDA, Farias MS, Barbosa E, Bresolin NL, Mehta NM, Moreno YMF. Enteral Protein Supplementation in Critically Ill Children: A Randomized Controlled Pilot and Feasibility Study. JPEN J Parenter Enteral Nutr. 2019 Feb;43(2):281-289. doi: 10.1002/jpen.1416. Epub 2018 Jun 30. PMID 29959852
- [Background] Mehta NM, Bechard LJ, Zurakowski D, Duggan CP, Heyland DK. Adequate enteral protein intake is inversely associated with 60-d mortality in critically ill children: a multicenter, prospective, cohort study. Am J Clin Nutr. 2015 Jul;102(1):199-206. doi: 10.3945/ajcn.114.104893. Epub 2015 May 13. PMID 25971721
- [Background] Wieczorek B, Ascenzi J, Kim Y, Lenker H, Potter C, Shata NJ, Mitchell L, Haut C, Berkowitz I, Pidcock F, Hoch J, Malamed C, Kravitz T, Kudchadkar SR. PICU Up!: Impact of a Quality Improvement Intervention to Promote Early Mobilization in Critically Ill Children. Pediatr Crit Care Med. 2016 Dec;17(12):e559-e566. doi: 10.1097/PCC.0000000000000983. PMID 27759596
- [Background] Choong K, Canci F, Clark H, Hopkins RO, Kudchadkar SR, Lati J, Morrow B, Neu C, Wieczorek B, Zebuhr C. Practice Recommendations for Early Mobilization in Critically Ill Children. J Pediatr Intensive Care. 2018 Mar;7(1):14-26. doi: 10.1055/s-0037-1601424. Epub 2017 Apr 10. PMID 31073462